CLINICAL TRIAL: NCT03924141
Title: Effects of a Brief De-escalation Training Program on Student Nurses' Skills and Confidence Level in Coping With Patient Aggression: a Cluster Randomized Controlled Study
Brief Title: Evaluation of Training in De-escalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bergen University College (Other)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Principal Investigator, Thomas Nag, Advisor, Bergen University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 716537
Record Dates: First submitted 2019-04-10; First posted 2019-04-23 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: De-escalation Skills
Keywords: De-escalation; Aggression; Violence prevention
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors who will assess the video data will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Third year nursing students - intervention (Experimental): Third year nursing students will receive the intervention in de-escalation training
  Interventions: Behavioral: Training in de-escalation
- Third year nursing students - control (No Intervention): Third year nursing students will receive no training in de-escalation

INTERVENTIONS:
Behavioral: Training in de-escalation — Will receive one hour of de-escalation training
  Arms: Third year nursing students - intervention

SUMMARY:
The purpose of the study is to evaluate one of the chapters in the new national Norwegian training manual (MAP). The chapter that is selected to be evaluated is the chapter on de-escalation. Effective training in this topic should not only lead to changes in the level of knowledge and attitudes, but also changes in behavior and skills. Experiencing better preparedness does not necessarily entail a change in behavior. This study wants to test whether training in de-escalation changes the participants' skills and experience of self-confidence, security and coping in threatening situations.

DETAILED DESCRIPTION:
The theme is:

• Evaluation of the training program of de-escalation for third-year nursing students

Underlying research questions will be:

* Will the intervention provide increased de-escalation skills?
* Will training in de-escalation provide increased confidence in coping with patient aggression?

The design used to answer the research questions is a cluster-randomized controlled study with an intervention group and a control group.

The two study groups with nursing students will be exposed to two different scenarios (A and B) with simulated patient situations. Students will conduct simulation A before the intervention and simulation B the same day after the intervention. A control group will also be included which will review scenarios A and B without intervention. The purpose of this is to see if the scenarios in isolation give any effect on the pre- and post-measurements.

Participants will also be asked to complete a questionnaire (Thackreys, 1987) related to experienced coping security related to aggression management at four different times.

The scenarios will be recorded on video. Following all video data collection, 2 de-escalation experts will independently review the video data and quantify it using the EMDABS instrument. They will be blinded and not aware of whether the video was recorded before or after the intervention. The data that this generates will then be statistically examined.

The selection of participants will be made from three classes with third year nursing students. The classes consist of about 50 students. Participation is voluntary.

It is uncertain how many will participate, but on the basis of practical limits there is an upper limit of 15 participants per class for the intervention group (the selection is recruited from two classes), and 30 participants from the control group (the selection is recruited from a class). A total of n = 30 is desired in both the intervention group and the control group.

The following two outcomes will be analyzed; de-escalating behavior (EMDABS, Mavandadi et al., 2016) and confidence in coping with patient aggression (Thackrey, 1987).

ELIGIBILITY:
Inclusion Criteria:

* Third year nursing student

Exclusion Criteria:

* Has to talk and understand Norwegian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in de-escalation skills: Baseline | Immediately before and immediately after intervention (single day, baseline)
  Instrument: "English Modified De-escalating Aggressive Behaviour Scale" (Mavandadi & Bieling, 2016)
Changes in de-escalation skills | Immediately before and immediately after intervention (single day, 6 months post-baseline)
  Instrument: "English Modified De-escalating Aggressive Behaviour Scale" (Mavandadi & Bieling, 2016)
Changes in de-escalation skills | Immediately before and immediately after intervention (single day, 9 months post-baseline)
  Instrument: "English Modified De-escalating Aggressive Behaviour Scale" (Mavandadi & Bieling, 2016)

SECONDARY OUTCOMES:
Changes in coping and confidence | Immediately before and immediately after intervention (single day, baseline)
  Instrument: "Clinicians confidence in coping with patient aggression" (Thackreys, 1987)
Changes in coping and confidence | Immediately before and immediately after intervention (single day, 6 months post-baseline)
  Instrument: "Clinicians confidence in coping with patient aggression" (Thackreys, 1987)
Changes in coping and confidence | Immediately before and immediately after intervention (single day, 9 months post-baseline)
  Instrument: "Clinicians confidence in coping with patient aggression" (Thackreys, 1987)

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Alsaker, PhD, Study Chair — Bergen University College
Locations (1):
- Bergen University College, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No